CLINICAL TRIAL: NCT05416450
Title: Comparison of the Efficacy of Intravaginal Electrical Stimulation in Antimuscarinic Naive and Refractory Women With Idiopathic Overactive Bladder
Brief Title: The Efficacy of Intravaginal Electrical Stimulation in Women With Idiopathic Overactive Bladder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Necmettin Yildiz, Clinical Professor, Pamukkale University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PamukkaleU-Unal-001
Record Dates: First submitted 2022-06-08; First posted 2022-06-13 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Urinary Bladder, Overactive
Keywords: bladder training; intravaginal electrical stimulation
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Antimuscarinic Naive (AM-N) (Active Comparator): None of the women had previously taken anti-muscarinic agents and oral ß3 adrenoreceptor agonist (mirabegron) in this group.
  Interventions: Device: intravaginal electrical stimulation added to bladder training
- Antimuscarinic Refractory (AM-R) (Active Comparator): Women with idiopathic OAB refractory to anti-muscarinic agents and oral ß3 adrenoreceptor agonist (mirabegron) when 2 or more were administered for at least 6 weeks each and failure was due to lack of efficacy with or without side effects were included in this group.
  Interventions: Device: intravaginal electrical stimulation added to bladder training

INTERVENTIONS:
Device: intravaginal electrical stimulation added to bladder training — BT was given as a home program. After information session, squeezing the PFM was shown in practice at least once to use in the urgency suppression strategies via digital palpation technique. The second stage strategies was aimed to delay urination, inhibit detrusor contraction, and prevent urgency by squeezing the PFM several times on a row, breathing deeply and self-motivating. In the third stage, a timed voiding program was started; a timed voiding and increasing the time between urination considering the voiding diary. IVES was applied in addition to BT in both groups. It was performed in lithotomy position via a stimulation device (Enraf Nonius Myomed 632) with a vaginal probe; three days a week, a total of 24 sessions for 8 weeks. Every session lasted 20 minutes. The stimulation parameters were a 10 Hz of frequency, a 5-10 s of work-rest cycle duration and, a 100 ms of pulse width. The symmetric biphasic pulse wave could be delivered over a range of 1-100 mA.

SUMMARY:
In this study, it was aimed to compare the effectiveness of intravaginal electrical stimulation (IVES) added to bladder training (BT) on quality of life (QoL) and clinical parameters related to overactive bladder (OAB) in antimuscarinic naive and refractory women. The results of this study would make it easier to understand the place of IVES among the treatment options in women with idiopathic OAB.

DETAILED DESCRIPTION:
Overactive bladder (OAB) is a symptom complex defined as urgency, with or without urgency urinary incontinence (UUI), usually with frequency and nocturia in the absence of urinary tract infection. Some authors listed the treatment options in idiopathic OAB as follows; first-line - behavioral therapy (lifestyle modifications, pelvic floor muscle (PFM) training, bladder training (BT), timed voiding), second-line - pharmacologic (antimuscarinic, beta-3 agonists), and third-line - neuromodulation/chemodenervation (tibial nerve stimulation, sacral neuromodulation, intradetrusor botulinum toxin). Intravaginal electrical stimulation (IVES) is involved in pelvic floor muscle training as a first-line treatment option. On the contrary, some authors stated that "the first-line treatment of idiopathic OAB includes behavior modification and physical therapy, and neuromodulation methods are used as third-line therapy in cases refractory to first-line and second-line (pharmacological) treatment. IVES, tibial nerve stimulation, and sacral neuromodulation are included as neuromodulation options". However, it is known that many patients with idiopathic OAB receive pharmacological treatment before reaching a conservative treatment option such as IVES. In common practice, antimuscarinic agents are frequently used as an initial treatment although burdened by a low adherence, and these patients need protracted treatment with periodic controls.

Some studies included subjects were not used antimuscarinics within the last 4-12 weeks or antimuscarinic-naive patients with OAB, while some included patients with OAB who were unresponsive or intolerant to antimuscarinics. As a result, IVES appear to be effective therapies used both as first-line treatment, as well as in managing refractory patients with idiopathic OAB. There is no evidence that it is most effective in which patients (antimuscarinic naive and refractory). Would it be more effective on the first-line or the third-line? or in other words; is there a difference in response to IVES in antimuscarinic naive and refractory patients with OAB? It should be kept in mind that IVES may lead to different results in antimuscarinic naive and refractory patients with idiopathic OAB. This study is the first prospective trial that compares the efficacy of IVES in antimuscarinic naive and refractory women with idiopathic OAB. In this study, it was aimed to compare the effectiveness of IVES added to BT on quality of life (QoL) and clinical parameters related to OAB in antimuscarinic naive and refractory women. The results of this study would make it easier to understand the place of IVES among the treatment options in women with idiopathic OAB.

ELIGIBILITY:
Inclusion Criteria:

* Over the age of 18 with the clinical diagnosis of idiopathic OAB
* Who could able to give written informed consent and understand the procedures

Exclusion Criteria:

* Women who had stress urinary incontinence
* A history of conservative therapy (BT, ES) for OAB within 6 months
* Urogynecological surgery within 3 months
* Current vulvovaginitis or urinary tract infections or malignancy
* Pregnancy
* Cardiac pacemaker or implanted defibrillator
* Anatomic structural disorders of the genital region that did not allow to apply the vaginal probe
* The strength of PFM less than 3/5 (graded as modified Oxford scale, min:0-max:5)
* The pelvic organ prolapse quantification (POP-Q) (stage 2 or more)
* Neurogenic bladder
* The peripheral or central neurologic pathology
* Ultrasonographic evidence of post-void residual urine volume more than 100 ml
* Allergy to condom or lubricant gel that is used with vaginal probe

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2022-12-15 (Estimated); Study Completion 2023-01-05 (Estimated)

PRIMARY OUTCOMES:
Incontinence episodes (positive response rate) | Change from baseline at the 8th week after the treatment
  To determine positive response rate, reduction in incontinence episodes was collected from the 3-day bladder diary. Women with ≥a 50% reduction in incontinence episodes were considered positive responders.

SECONDARY OUTCOMES:
the severity of incontinence | Change from baseline at the 8th week after the treatment
  The 24-hour pad test was carried out to evaluate the severity of incontinence .
symptom severity | Change from baseline at the 8th week after the treatment
  Overactive Bladder Questionnaire (OAB-V8) was used to evaluate the symptom severity in patients with OAB in this study. The OAB-V8 consists of 8 questions in which the patients can be classified with respect to the symptom severity: none (0), very little (1), a little (2), quite a few (3), very (4), and too many (5). The total score ranges from 0-40.
frequency of voiding | Change from baseline at the 8th week after the treatment
  The frequencies of voiding, nocturia, and the number of pads used were collected from the 3-day bladder diary.
nocturia | Change from baseline at the 8th week after the treatment
  The frequencies of voiding, nocturia, and the number of pads used were collected from the 3-day bladder diary.
number of pads | Change from baseline at the 8th week after the treatment
  The frequencies of voiding, nocturia, and the number of pads used were collected from the 3-day bladder diary.
quality of life (QoL) | Change from baseline at the 8th week after the treatment
  The Quality of Life-Incontinence Impact Questionnaire (IIQ7) was used to assess specific QoL related to incontinence. Minimum score is 0, maximum score is 21 and high scores mention worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Necmettin Yıldız, Prof, Study Director — Pamukkale University
Locations (1):
- Pamukkale Univercity, Denizli, Turkey (Türkiye)

REFERENCES:
- [Derived] Yildiz N, Unal B. Comparison of the efficacy of intravaginal electrical stimulation in women with idiopathic overactive bladder naive and refractory to pharmacological agents. Int Urogynecol J. 2023 Sep;34(9):2099-2105. doi: 10.1007/s00192-023-05517-1. Epub 2023 Mar 28. PMID 36976326